CLINICAL TRIAL: NCT06473571
Title: Testing a Strategy to Improve the Effects of Caregiving for Caregivers of Persons with Dementia
Brief Title: Effects on Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004299
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Dementia
Keywords: dementia; caregivers
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Protocol (The 3GT) (Active Comparator): Participants will be asked to identify three things that went well that day and their role for this occurring ["What went well today, and what was your role in making it happen?" as adapted from (Sexton & Adair, 2019)]. They will be asked to engage in this exercise for 15 days during the evening.
  Interventions: Other: Intervention Protocol (The 3GT)
- Control Group (Active Comparator): Participants will be asked to reflect on early memories of their life, with no specific prompts provided, for 15 days during the evening. This activity is consistent with prior efficacy studies of 3GT (Seligman et al., 2005).
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Protocol (The 3GT) — Participants will be asked to identify three things that went well that day and their role for this occurring ["What went well today, and what was your role in making it happen?" as adapted from (Sexton & Adair, 2019)]. They will be asked to engage in this exercise for 15 days during the evening.
  Arms: Intervention Protocol (The 3GT)
Other: Control Group — Participants will be asked to reflect on early memories of their life, with no specific prompts provided, for 15 days during the evening. This activity is consistent with prior efficacy studies of 3GT (Seligman et al., 2005).
  Arms: Control Group

SUMMARY:
The Three Good Things (3GT) is a gratitude list intervention that is empirically supported (Emmons & McCullough, 2003; Seligman et al., 2005) and is a low-cost, easily accessible tool for medical and mental providers to recommend and dementia caregivers to implement independently. Thus, this study aims to investigate the feasibility of use of 3GT in the dementia caregiving population and investigate potential therapeutic mechanisms of the intervention.

DETAILED DESCRIPTION:
The hypothesis predicts that Caregivers of persons diagnosed with dementia who are randomized into the intervention group (3GT) will report reduced levels of depression, burden, burnout, show an increase in levels of gratitude, increased positive emotion, and increased positive reframing (Brief COPE: Positive Reinterpretation scale and Positive Aspects of Caregiving measure) as compared to baseline levels, and post-follow up assessment in 15 days. The participants will be recruited from local community partners and Amazon MTurk. They will be randomized into 2 groups; one group will be asked to reflect on three good things that happened that day, and the other group will be asked to reflect on early memories. Participants will be reminded via text message daily for 15 days and asked to document their three good things or early memories on a Qualtrics link that will be provided in the text message. Additionally, they will be asked to answer 10 mood-related questions daily. An ANOVA will be used to assess the pre and post intervention differences between groups for depression, burden, burnout, gratitude, positive emotion, and positive reframing. Multilevel modeling will be used to assess the relationships between gratitude and depression at the within-subjects level and then between-subjects by intervention condition. Identified demographic factors will be added to covary at both levels of analysis. Data will be de-identified and stored on a University of Central Florida local hard drive, which requires special permission and password-protected profiles.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified caregivers of persons with dementia at least 18 years of age
* Identify English as their primary language
* Self-report current care for an older adult with dementia identified by a medical professional

Exclusion Criteria:

* Participants that are currently receiving psychotherapy, have a diagnosis of dementia, and/or severe mental illness
* Individuals under the age of 18 years old
* Adults who cannot consent in English
* Pregnant women and prisoners will not be included in the study.
* Participants who do not have access to a phone that can not receive text messages will not be able to participate, as equipment will not be provided to Participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
To measure gratitude using The Gratitude Questionnaire (GQ-6) | 6 months
  The Gratitude Questionnaire (GQ-6), which is a widely used measure trait gratitude will be used. The GQ-6 is a 6 item self-report questionnaire that assesses gratitude disposition in an individual.
To measure depressive symptoms using the Center for Epidemiologic Studies Depression Scale (CES-D 10) | 6 months
  For this study, the 10-item Center for Epidemiologic Studies Depression Scale (CES-D 10) will be used to measure depressive symptoms
To measure burnout using The Informal Caregiver Burnout Inventory 10 (ICBI-10) | 6 months
  The Informal Caregiver Burnout Inventory 10 (ICBI-10) is a new measure developed to capture burnout specifically in caregivers, aiming to validate prior attempts to modify language in general use burnout measures that typically capture occupational burnout.
To assess positive emotion using The Positive and Negative Affect Schedule (PANAS) | 6 months
  The Positive and Negative Affect Schedule (PANAS) will be utilized to assess positive affect. The PANAS is a 20-item self-report measure assessing two dimensions of affect (positive and negative) utilizing 5-point Likert scale.
To measure positive reframing using the Brief COPE Inventory: Positive Reinterpretation subscale | 6 months
  To measure positive reframing, the Brief COPE Inventory: Positive Reinterpretation subscale will be used (Items 12 and 17), which is a measure that assess different types of coping utilized by individuals in stressful situations.
To evaluate practical implications of positive reframing using the Positive Aspects of Caregiving measure | 6 months
  The Positive Aspects of Caregiving measure is a 9-item self-report scale assessing the positive factors associated with caregiving, utilizing a 5-point Likert scale ranging from 1 ("Disagree a lot") to 5 ("Agree").
Assess caregiver burden using the Zarit Burden Interview | 6 months
  The Zarit Burden Interview, short form (ZBI-SF) will be used to measure participants subjective burden related to their caregiving role.
To asses ICN1-10 validity, the Burnout Measure, Short (BMS) will be used | 6 months
  To provide convergent validity for the use of the ICBI-10 in this sample, the Burnout Measure, Short (BMS) will be used, which is a widely used measure of burnout. The BMS is a 10-item, self-report measure that assess three factors of burnout including physical, emotional and mental exhaustion.
To measure daily depressive symptoms using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) | 6 months
  4 questions adapted from the The NIH Patient-Reported Outcomes Measurement Information System (PROMIS) short form depression item will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole McClure, MS, MA, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States